CLINICAL TRIAL: NCT01567397
Title: Registry of Dupuytren's Contracture Treatment Outcomes
Acronym: ReDuCTO
Status: Completed | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Collaborators: GWT-TUD GmbH (Other); Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: ReDuCTO ID 7090
Record Dates: First submitted 2012-03-28; First posted 2012-03-30 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Dupuytren's Disease
MeSH Terms: conditions — Dupuytren Contracture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Experience with Microbial Collagenase (trade name Xiapex) in Europe currently is limited to randomised controlled studies.While such studies are essential to determine efficacy and safety of the product (usually compared to placebo), they provide no information on the effectiveness of the drug and further aspects of its use (feasibility, tolerability, quality of life and other patient-related outcomes) in the typical "real-life" setting under clinical practice conditions.Thus, the present study aims to collect data on the

* Drug utilization of Microbial Collagenase in the hand of physicians, with focus on feasibility, treatment patterns, and effectiveness in clinical practice
* Context of Microbial Collagenase therapy (setting, patient characteristics, concomitant treatment, follow-up therapy)
* Effectiveness (with focus on functionality)
* Tolerability
* Patient-related outcomes: patient satisfaction, health-related quality of life
* Physician satisfaction with therapy
* Resource utilization (hospital stays, drug consumption, concomitant medication etc.)
* Long-term outcomes

ELIGIBILITY:
Inclusion Criteria:

* palpable cord due to Dupuytren's Disease (pretreated or untreated)
* satisfactory knowledge of German to be able to fill out questionnaires
* written informed consent

Exclusion Criteria:

* contraindication to Microbial Collagenase (according to Prescription Information)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Dupuytren's Disease
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2011-12; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Pittrow, MD, PhD, Study Director — Institute for Clinical Pharmacology, Medical Faculty, Technical University Dresden, Germany; Wilhelm Kirch, MD, PhD, Principal Investigator — Institute for Clinical Pharmacology (Director), Medical Faculty, Technical University, Dresden, Germany; Max Härle, MD, Study Director — Orthopädische Klinik, Markgröningen, Germany; Jörg Witthaut, MD, Study Director — Schön Klinik Vogtareuth; Riccardo Giunta, MD, Study Director — Hand Surgery, Ludwig-Maximilian-University Munich, Germany
Locations (4):
- Germany (4):
  - Prof. Dr. Max Haerle, Markgröningen
  - Prof. Dr. Riccardo Giunta, Munich
  - Several undisclosed sites, Various Cities
  - Dr. Joerg Witthaut, Vogtareuth

REFERENCES:
- See also: Publication of results in the German Mecial Science (GMS) database — http://www.egms.de/static/de/journals/gpras/2015-5/gpras000034.shtml